CLINICAL TRIAL: NCT00305799
Title: Auditory and Vestibular Function Evaluation in Patients With Solid Tumors Treated With Oxaliplatin-Containing Chemotherapy
Brief Title: Hearing Loss and Dizziness in Patients Receiving Oxaliplatin for Solid Tumors
Status: Completed | Type: Observational
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CASE3Y05; P30CA043703 (NIH); CASE3Y05 (Other: Case Comprehensive Cancer Center); 10-05-19 (Other: University Hospitals IRB)
Record Dates: First submitted 2006-03-21; First posted 2006-03-22 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-11

CONDITIONS: Neurotoxicity; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: neurotoxicity; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Neurotoxicity Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: management of therapy complications — Patients will complete three self-reported questionnaires including the Peripheral Neuropathy Scale, Hearing Handicap Inventory for Adults, and Dizziness Handicap Inventory. Patients will also be asked a series of questions regarding symptoms or complaints about hearing changes, tinnitus, and dizziness that they may have experienced prior to, during, and after completion of chemotherapy. Patients will also undergo a hearing test.

SUMMARY:
RATIONALE: Understanding how oxaliplatin affects hearing loss, dizziness, and peripheral neuropathy may improve the ability to plan effective treatment for patients receiving oxaliplatin for solid tumors.

PURPOSE: This clinical trial is studying hearing loss and dizziness in patients receiving oxaliplatin for solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Define the prevalence of audiometrically detectable hearing loss in patients with solid tumors treated with oxaliplatin.
* Describe the association of chemotherapy-induced peripheral neuropathy (CIPN) and audiometrically detectable hearing loss in these patients.
* Describe the association of CIPN and patient self-reported scales including, Peripheral Neuropathy Scale, Hearing Handicap Inventory for Adults, and Dizziness Handicap Inventory.

OUTLINE: This is an exploratory study.

Patients will complete three self-reported questionnaires including the Peripheral Neuropathy Scale, Hearing Handicap Inventory for Adults, and Dizziness Handicap Inventory. Patients will also be asked a series of questions regarding symptoms or complaints about hearing changes, tinnitus, and dizziness that they may have experienced prior to, during, and after completion of chemotherapy. Patients will also undergo a hearing test.

PROJECTED ACCRUAL: A total of 60 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of solid tumor

  * Received an oxaliplatin-containing chemotherapy regimen within the past 15 months* NOTE: *If oxaliplatin was omitted from the patient's most recent chemotherapy regimen due to ototoxicity, the patient is still eligible for participation in this study
* No known CNS metastases

PATIENT CHARACTERISTICS:

* No history of spinal injuries
* ECOG performance status 0-3
* No history of chronic renal failure
* No known HIV/AIDS

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2005-11; Primary Completion 2012-12 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Hearing loss as measured by Hearing Loss Inventory, Dizziness Handicap Inventory, and audiogram every 2 months during treatment, and then 2-4 weeks and 6 months after completion of study treatment | every 2 months during treatment, and then 2-4 weeks and 6 months after completion of study treatment
Peripheral neuropathy as measured by Peripheral Neuropathy Scale every 2 months during treatment, and then 2-4 weeks and 6 months after completion of study treatment | every 2 months during treatment, and then 2-4 weeks and 6 months after completion of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sabarish Ayyappan, MD, Study Chair — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio